CLINICAL TRIAL: NCT06112054
Title: Impedance Sensor Evaluated in Peripheral Artery Disease for Tissue Detection
Acronym: SEPARATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sensome (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SEN-PAD-1
Record Dates: First submitted 2023-10-15; First posted 2023-11-01 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Peripheral Vascular Disease
Keywords: PAD
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Intervention Model Description: Single center, single group, non comparative study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): One arm only - in all eligible study patients, the study device will be used.
  Interventions: Device: Clotild Smart Guidewire System (CSGS)

INTERVENTIONS:
Device: Clotild Smart Guidewire System (CSGS) — In the current study, a commercially available CE marked guidewire will be used to direct a catheter through blood vessels while the Clotild® Smart Guidewire (study device) will only be used to perform electrophysiological measurements (via its sensors) in the blood vessels during peripheral endovascular procedures. It is thus designed for use as an adjunct to conventional angiographic procedure

SUMMARY:
The objective of the study is to evaluate the feasibility of the CSGS sensor to differentiate tissues involved in Peripheral Artery Disease (PAD).

DETAILED DESCRIPTION:
The objective of the study is to evaluate the feasibility of the CSGS sensor to differentiate tissues involved in Peripheral Artery Disease (PAD)

Previously the CSGS was used in a clinical study in stroke patients (The Clot Out Study) to direct a catheter through blood vessels and to measure electrophysiological parameters in the blood vessels during procedures.

In the current study however, a commercially available CE marked guidewire will be used to direct a catheter through blood vessels while the Clotild® Smart Guidewire System will only be used to perform electrophysiological measurements in the blood vessels during peripheral endovascular procedures. It is thus designed for use as an adjunct to conventional angiographic procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Subjects with acute and chronic occlusions in the arteries of the lower limbs
* Patients eligible for endovascular interventional procedures
* Written Informed Consent to participate in the study.

Exclusion Criteria:

* Target Vessel Aneurysm
* Target vessel diameter <2mm
* Lesions starting at the Common Iliac Artery
* Any subject that is, according to the discretion of the investigator, not eligible for study participation
* Known lactating or confirmation of positive pregnancy test according to site specific standard of care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2024-08-14 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
The ability of Clotild® Smart Guidewire System to acquire electrophysiological measurements in the lesion and/or subintimal. | During the procedure
  The Primary Performance Endpoint is defined as the ability of Clotild® Smart Guidewire System to acquire electrophysiological measurements in the lesion and/or subintimal. Data of the 9 individual impedance measurements will be collected during the procedure and might be aggregated at the row level or sensor level. This endpoint represents the procedural success rate being defined as the CSGS obtaining at least one non-anomalous impedance measurement in the lesion during the procedure.

SECONDARY OUTCOMES:
The ability of Clotild® Smart Guidewire System to differentiate various tissues involved in Peripheral Artery Disease | During the procedure
  The ability of Clotild® Smart Guidewire System to differentiate various tissues involved in Peripheral Artery Disease such as, but not limited to: • arterial wall
  * subintimal area
  * clot (fresh / subacute / organised)
  * plaque (soft / hard)
  * hyperplasia
  The ability to differentiate tissues will be reported by descriptive statistics.
  To further assess the secondary endpoint, Machine Learning analysis will be applied. Following standard procedure, features will be extracted from the impedance measurements and used for model inference.

CONTACTS AND LOCATIONS:
Locations (1):
- AZ Sint Blasius, Dendermonde, Belgium

IPD SHARING:
Plan to Share IPD: No